CLINICAL TRIAL: NCT03191812
Title: Optimization of Transcranial Direct Current Stimulation (tDCS) for Dual Task Performance in Older Adults With and Without a History of Falls
Brief Title: The Short-term Effects of Noninvasive Electrical Brain Stimulation on Dual Tasking in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Brad Manor, Associate Scientist, Hebrew SeniorLife
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2016-26
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Aging
Keywords: Falls; transcranial Direct Current Stimulation; Mobility; Dual Task
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sham Stimulation (Sham Comparator): The Sham stimulation intervention will consist of one, twenty-minute session of transcranial direct current stimulation (tDCS) that does not target a cortical area but instead, provides just enough current to create tingling sensations across the scalp to mimic the feeling of receiving the real stimulation. The sham stimulation will use the same number and placement of electrodes as the real stimulation but with a much smaller total current intensity of 0.5 milliamps (mA).
  Interventions: Other: transcranial Direct Current Stimulation (tDCS)
- M1 Stimulation (Experimental): The M1 stimulation intervention consists of one, twenty-minute session of transcranial direct current stimulation (tDCS) targeting the primary motor cortex at a total current intensity of 1.5 mA.
  Interventions: Other: transcranial Direct Current Stimulation (tDCS)
- DLPFC Stimulation (Experimental): The DLPFC stimulation intervention consists of one, twenty-minute session of transcranial direct current stimulation (tDCS) targeting the dorsolateral prefrontal cortex at a total current intensity of 1.5 mA.
  Interventions: Other: transcranial Direct Current Stimulation (tDCS)
- M1+DLPFC Stimulation (Experimental): The M1+DLPFC stimulation intervention consists of one, twenty-minute session of transcranial direct current stimulation (tDCS) targeting the primary motor cortex and the dorsolateral prefrontal cortex simultaneously at a total current intensity of 3.0 mA.
  Interventions: Other: transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Other: transcranial Direct Current Stimulation (tDCS) — There will be three different tDCS targets as well as a sham stimulation condition. The stimulation for each of these conditions will be delivered via 6 already-placed gel electrodes on the participant's scalp with different combinations of current intensities among all the electrodes.

SUMMARY:
The tDCS & Dual Tasking study will compare the effects of transcranial Direct Current Stimulation (tDCS) targeting three different cortical regions (as well as sham stimulation) on dual task standing and walking in older adults with and without a recent history of recurrent falls.

DETAILED DESCRIPTION:
The ability to stand and walk safely, especially while performing additional cognitive tasks like talking, reading or decision making, is critical to the preservation of functional independence into old age. Such "dual tasking" often impairs balance, even in healthy older adults and those with greater dual task "costs" are more likely to suffer future falls. Transcranial direct current stimulation (tDCS) is a safe, noninvasive and inexpensive means of modulating activity across cortical networks. A single, 20-minute session of tDCS facilitates brain activity for up to 24 hours. Through Dr. Manor's previous research in healthy older adults, he has discovered that just 20 minutes of tDCS targeting the left dorsolateral prefrontal cortex (dlPFC)-a region involved in both cognitive and motor function-immediately reduces the dual task costs to balance when standing and walking, and improves performance in the timed up-and-go (TUG) test of mobility. However, there are several brain networks with known involvement in balance control and dual tasking, and the optimal brain region to target to improve dual task capacity has not been established. The proposed study will be a double-blinded, sham-controlled study in which older adults both with and without a history of falling undergo dual task assessments immediately before and after single, 20-minute sessions of tDCS designed to target several different brain regions with known involvement in dual tasking and the maintenance of balance.

ELIGIBILITY:
Inclusion Criteria:

"Faller" group

* Aged 65 years and older
* Able to read, write and communicate in English
* Self-report of 2 or more falls within the past 6 months

"Non-Faller" Group

* Aged 65 years and older
* Able to read, write, and communicate in English
* Self-report of 1 or no (zero) falls within the past 6 months

Exclusion Criteria:

* Self-reported diagnosis of Parkinson's disease, Alzheimer's disease or dementia, multiple sclerosis, history of stroke or other neurodegenerative disorder.
* Self-reported active cancer for which chemo-/radiation therapy is being received.
* Hospitalization within the past 3 months due to acute illness or as a result of a musculoskeletal injury significantly affecting gait and balance.
* Montreal Cognitive Assessment score <18, or insufficient understanding of study procedures following review of the Informed Consent Form. Understanding will be assessed by asking the participant to answer the following three questions: 1) What is the purpose of this study? 2) What are the risks of study involvement? 3) If you decide to participate, are you allowed to withdraw from the study at any time? Answers will be recorded by study personnel on the "Assessment of Protocol Understanding" form (see attached). Insufficient understanding will be defined by one or more incorrect answers, as determined at the discretion of the investigator.
* Inability to stand or ambulate unassisted for at least 25 feet.
* Contraindications to tDCS, including a reported seizure within the past two years, use of neuro-active drugs, the risk of metal objects in the brain, skull, or head, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant), or the presence of any active dermatological condition, such as eczema, on the scalp (see appendix for standardized tDCS screening questionnaire).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Dual task cost to standing postural sway speed | This outcome will be assessed immediately before and after each 20-minute session of tDCS.
  The dual task cost to standing postural sway speed will be calculated from trials of standing with and without simultaneous performance of a serial subtraction cognitive task. The dual task cost will be calculated as the percent change in sway speed from single- to dual-task conditions.
Dual task cost to gait speed when walking | This outcome will be assessed immediately before and after each 20-minute session of tDCS.
  The dual task cost to gait speed when walking will be calculated from trials of walking with and without simultaneous performance of a serial subtraction cognitive task. The dual task cost will be calculated as the percent change in gait speed from single- to dual-task conditions.

SECONDARY OUTCOMES:
Dual task cost to postural sway area | This outcome will be assessed immediately before and after each 20-minute session of tDCS.
  The dual task cost to standing postural sway area will be calculated from trials of standing with and without simultaneous performance of a serial subtraction cognitive task. The dual task cost will be calculated as the percent change in postural sway area from single- to dual-task conditions.
Dual task cost to gait variability when walking | This outcome will be assessed immediately before and after each 20-minute session of tDCS.
  The dual task cost to gait variability when walking will be calculated from trials of walking with and without simultaneous performance of a serial subtraction cognitive task. Gait variability will be defined as the coefficient of variation about the average stride time (stride times defined by the time between consecutive heel strides of the same leg). The dual task cost will be calculated as the percent change in gait variability from single- to dual-task conditions.
Single task postural sway speed | This outcome will be assessed immediately before and after each 20-minute session of tDCS.
  Single task postural sway speed will be calculated from trials of standing without simultaneous performance of a serial subtraction cognitive task.
Single task postural sway area | This outcome will be assessed immediately before and after each 20-minute session of tDCS.
  Single task postural sway area will be calculated from trials of standing without simultaneous performance of a serial subtraction cognitive task.
Single task gait speed variability when walking | This outcome will be assessed immediately before and after each 20-minute session of tDCS.
  Single task gait variability when walking will be calculated from trials of walking without simultaneous performance of a serial subtraction cognitive task. Gait variability will be defined as the coefficient of variation about the average stride time (stride times defined by the time between consecutive heel strides of the same leg).
Single task gait speed when walking | This outcome will be assessed immediately before and after each 20-minute session of tDCS.
  Single task gait speed when walking will be calculated from trials of walking without simultaneous performance of a serial subtraction cognitive task.
Mobility | This outcome will be assessed immediately before and after each 20-minute session of tDCS.
  Mobility will be assessed using the Timed Up-and-Go test in which the amount of time it takes for the participant to stand up from a chair, walk three meters, turn around a cone, walk back, and sit down is recorded.
Executive function | This outcome will be assessed immediately before and after each 20-minute session of tDCS.
  Executive function will be assessed using the Stroop test.
Cognitive processing speed | This outcome will be assessed immediately before and after each 20-minute session of tDCS.
  Cognitive processing speed will be assessed using the Symbol Digit Modalities Test (SDMT).
Attention | This outcome will be assessed immediately before and after each 20-minute session of tDCS
  Attention will be assessed using the Visual Search and Attention Test (VSAT).

CONTACTS AND LOCATIONS:
Overall Officials: Brad Manor, Principal Investigator — Institute for Aging Research, Hebrew SeniorLife
Locations (2):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States
- Laboratory for Gait and Neurodynamics, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No